CLINICAL TRIAL: NCT06079853
Title: The Use of Physiologic Measures and Sleep Health Promotion to Identify and Mitigate Predisposing Factors of Suicidal Ideation in Nurses
Brief Title: Nurse Suicide: Physiologic Sleep Health Promotion Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Allison Norful, Assistant Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU3204
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Suicide; Nurse's Role; Work Environment Adverse Effects; Sleep; Stress; Mental Health Wellness 1
Keywords: Suicide; Nurse; Sleep; Mental Health; Work Environment; Stress; Depression; Anxiety
MeSH Terms: conditions — Suicide; Occupational Stress; Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Single arm pilot sample will receive intervention
  Interventions: Behavioral: PureSomni Sleep Health Product Kit

INTERVENTIONS:
Behavioral: PureSomni Sleep Health Product Kit — PureSomni sleep health products offered: blue light blocking glasses, eye mask, nasal strips, white noise machine, lavender spray, herbal tea, ear plugs

SUMMARY:
The purpose of this study is to identify factors (sleep, psychiatric characteristics, stressful life events, and work environment characteristics) that potentiate or mitigate adverse effects of real-world stressors that predispose nurses to suicidal risk.

The specific aims are:

Aim 1. To investigate associations between sleep, stressful life events (life stressors, discrimination, lateral violence), psychiatric characteristics (psychiatric diagnosis, subjective mood), work environment characteristics (workload, shift type and duration, overtime, nurse work environment, and team relations) and stress (self-report and heart rate variability) in working nursing professionals while controlling for standard covariates known to influence stress.

Aim 2. To determine if stress exposure (self-report and HRV) is associated with predisposing factors (sleep, stressful life events, additional psychiatric characteristics, and work environment characteristics), and to explore whether stress mediates the effect of predisposing factors on suicidal ideation in working nursing professionals.

Exploratory Aim. To explore the preliminary impact of an existing sleep intervention (sleep health promotion kit) on self-reported stress, HRV, sleep, and psychiatric health outcomes including depression, burnout, and suicidal ideation.

This record will focus on the Exploratory Aim.

DETAILED DESCRIPTION:
Despite being the largest healthcare workforce in the United States (US) (~5 million nurses), evidence about suicidal ideation and predisposing factors that contribute to suicide in nurses is limited. Outside of nursing, there is substantial evidence that an individual's psychiatric characteristics (psychiatric diagnosis; decision-making; social cognition; mood) and/or life stressors (e.g., death of a loved one, divorce, discrimination, or lateral violence) are significantly associated to suicidal ideation. Yet, it is unclear why nurses have higher rates of suicide compared to other populations and which factors predispose nurses to higher risk for suicidal behavior. It has become critical to test new approaches to reduce stress in nurses and subsequently mitigate suicide ideation. There is early evidence that sleep disturbances may induce increased stress and subsequently higher psychological risk, including depression, a known predisposing risk factor for suicidal risk. Evidence about the associations between sleep and suicidal ideation is limited but early studies show promise that interventions promoting sleep health may help mitigate suicidal risk. The isolation of predisposing factors for stress in nurses and investigation of potential interventions to counteract such stress may help to identify and mitigate suicide risk in nurses. Past evidence about suicide has been limited to post-mortem data inhibiting an understanding of which personal, psychosocial, and work environment factors predispose a nurse to suicidal behaviors. The combined study of self-report and physiologic data may help us better understand sources of stress adaptation in the search for underlying biological mechanisms associated with suicide and other suboptimal psychologic health outcomes.

ELIGIBILITY:
Inclusion criteria

* currently practicing as a registered nurse in the clinical setting
* have worked continuously in the same position for at least 1 year
* read, speak, and understand English language

Exclusion criteria

* >1-month sick leave in the past 3 months
* pregnancy (known physiologic stress confounder)
* other healthcare workers (e.g., physicians).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison A Norful, PhD, Principal Investigator — Columbia University School of Nursing
Locations (1):
- NewYork Presbyterian Hudson Valley Hospital, Cortlandt Manor, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Single arm participants will receive the intervention PureSomni Sleep Health Product Kit: blue light blocking glasses, eye mask, nasal strips, white noise machine, lavender spray, herbal tea, ear plugs
Period: Overall Study
Arm/Group | Experimental
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 25
Maslach Burnout Inventory (Subscale: Emotional Exhaustion) Baseline [Mean (Standard Deviation); unit: units on a scale] — Scaling - Self report survey (subscale 1-emotional exhaustion) 7 point Likert Scale; Score Range 0-42
  Interpretation:
  17 or less - Low level of burnout 18-29 - Moderate level of burnout Greater than 30 - High level of burnout
  units on a scale | 31.2 (11.72)
Maslach Burnout Inventory (Subscale: Depersonalization) Baseline [Mean (Standard Deviation); unit: units on a scale] — Scaling - Self report survey (subscale 2-Depersonalization) 7 point Likert Scale; Score Range 0-42
  Interpretation:
  5 or less - Low level of burnout 6-11 - Moderate level of burnout Greater than 12 - High level of burnout
  units on a scale | 10.84 (6.17)
Maslach Burnout Inventory (Subscale: Personal Accomplishment) Baseline [Mean (Standard Deviation); unit: units on a scale] — Scaling - Self report survey (subscale 3-Personal Achievement) 7 point Likert Scale; Score Range 0-48
  Interpretation:
  33 or less - Low level of burnout 34-39 - Moderate level of burnout Greater than 40 - High level of burnout
  units on a scale | 44.92 (7.49)

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Severity Rating Scale (Intensity of Ideation) - Number of Participants With a Positive CSSRS Ideation
Description: This outcome measures the number of participants who had a score greater than 0 on the CSSRS at Baseline (Week 1).
  CSSRS total score range is from 0-6, with the higher number indicating more intense ideation. Any score above 0 indicates a positive ideation in the past month.
Time Frame: Baseline: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 25
Participants | 2

2. Primary Outcome: Columbia Suicide Severity Rating Scale (Intensity of Ideation) - Number of Participants With a Positive CSSRS Ideation
Description: This outcome measures the number of participants who had a score greater than 0 on the CSSRS at Follow-up (Week 4).
  CSSRS total score range is from 0-6, with the higher number indicating more intense ideation. Any score above 0 indicates a positive ideation in the past month.
Time Frame: Follow-up: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 25
Participants | 0

3. Primary Outcome: Columbia Suicide Severity Rating Scale (Intensity of Ideation) - Number of Participants With a Positive CSSRS Ideation
Description: This outcome measures the number of participants who had a score greater than 0 on the CSSRS at Follow-up (Week 8).
  CSSRS total score range is from 0-6, with the higher number indicating more intense ideation. Any score above 0 indicates a positive ideation in the past month.
Time Frame: Follow-up: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 24
Participants | 0

4. Primary Outcome: Physiologic Stress Response- Heart Rate Variability [Group Mean Difference Between Week 1-4(Control) and Week 5-8(Intervention)]
Description: Participants will wear the OuraRing to capture physiologic continuous heart rate variability. Heart rate variability is the variance in time between heart beats (RR intervals on an EKG) and is calculated using root mean square of successive differences between heartbeats. The middle 50% of 20-25 year olds usually have an average HRV in the 55-105 range, while 60-65 year olds tend to be between 25-45. In general, a higher heart rate variability is considered better as it indicates a more adaptable and resilient autonomic nervous system, which can respond effectively to different stressors. We calculated the mean difference between the control time period (Week1-4) and the intervention time period (Week 5-8).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Experimental
Number analyzed (Participants) | 25
milliseconds | 0.846 (5.424)

5. Primary Outcome: Perceived Sleep Quality Via Pittsburgh Sleep Quality Index Global Sleep Score (Group Mean)
Description: Scaling: Self reported Survey Instrument Range: 0 to 21 Interpretation: A global sleep score over 5 indicates poor sleep quality.
Time Frame: baseline-Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 8.30 (3.91)

6. Primary Outcome: Perceived Sleep Quality Via Pittsburgh Sleep Quality Index Global Sleep Score (Group Mean)
Description: as for outcome 5
Time Frame: Follow up- Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 6.79 (3.37)

7. Primary Outcome: Perceived Sleep Quality Via Pittsburgh Sleep Quality Index Global Sleep Score (Group Mean)
Description: as for outcome 5
Time Frame: Follow up- Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 24
score on a scale | 5.85 (3.03)

8. Primary Outcome: Physiologic Sleep Data - Sleep Duration (Mean Daily Hours)
Description: This is to measure the average amount of daily sleep (hours) over an 8 week period. The physiologic data is collected via a wearable device (OuraRing).
  We calculated the mean difference in sleep duration (hours) between Week 1-4 (Control time period) and Week 5-8(Intervention time period).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Experimental
Number analyzed (Participants) | 24
Hours | 6.81 (0.831)

9. Primary Outcome: Number of Participants With at Least 1 Suicidal Behavior (Frequency)
Description: Total number of participants with at least 1 suicidal behavior that occurred during the given time period of 8 weeks.
Time Frame: 8 Weeks
Measure: Number; unit: participants
Arm/Group | Experimental
Number analyzed (Participants) | 25
participants | 0

10. Secondary Outcome: Burnout Screening Via Maslach Burnout Inventory (Subscale 1: Emotional Exhaustion) - Mean Composite Score
Description: Scaling - Self report survey (subscale 1-emotional exhaustion) 7 point Likert Scale; Score Range 0-42
  Interpretation:
  17 or less - Low level of burnout 18-29 - Moderate level of burnout Greater than 30 - High level of burnout
Time Frame: Baseline- Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 31.2 (11.72)

11. Secondary Outcome: Burnout Screening Via Maslach Burnout Inventory (Subscale 2: Depersonalization) - Mean Composite Score
Description: Scaling - Self report survey (subscale 2-Depersonalization) 7 point Likert Scale; Score Range 0-42
  Interpretation:
  5 or less - Low level of burnout 6-11 - Moderate level of burnout Greater than 12 - High level of burnout
Time Frame: Baseline- Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 10.84 (6.17)

12. Secondary Outcome: Burnout Screening Via Maslach Burnout Inventory (Subscale 3: Personal Accomplishment) - Mean Composite Score
Description: Scaling - Self report survey (subscale 3-Personal Achievement) 7 point Likert Scale; Score Range 0-48
  Interpretation:
  33 or less - Low level of burnout 34-39 - Moderate level of burnout Greater than 40 - High level of burnout
Time Frame: Baseline- Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 44.92 (7.49)

13. Secondary Outcome: Burnout Screening Via Maslach Burnout Inventory (Subscale 1: Emotional Exhaustion) - Mean Composite Score
Description: as for outcome 10
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 29 (14.4)

14. Secondary Outcome: Burnout Screening Via Maslach Burnout Inventory (Subscale 2: Depersonalization) - Mean Composite Score
Description: as for outcome 11
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 10.88 (5.69)

15. Secondary Outcome: Burnout Screening Via Maslach Burnout Inventory (Subscale 3: Personal Achievement) - Mean Composite Score
Description: as for outcome 12
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 25
score on a scale | 44.29 (9.5)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Sample Size is limited to pilot trial with 25 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT06079853/Prot_SAP_ICF_000.pdf